CLINICAL TRIAL: NCT00747630
Title: Evaluating the Efficacy of a Video Based Intervention to Educate Teen Moms About Fetal Alcohol Syndrome
Brief Title: Evaluating the Efficacy of a Video Based Intervention to Educate Teen Moms About Fetal Alcohol Syndrome (FAS)
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: This project was not a clinical trial requiring registration
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FAS Study
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Fetal Alcohol Syndrome; Teen Pregnancy
Keywords: Fetal Alcohol Syndrome; Teen pregnancy
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): The group selected to watch the video.
  Interventions: Other: An educational video about Fetal Alcohol Syndrome

INTERVENTIONS:
Other: An educational video about Fetal Alcohol Syndrome — A 20 minute video about FAS

SUMMARY:
Evaluating the efficacy of a video about FAS to determine whether it has an impact on knowledge about FAS and their likelihood to participate in risk taking behavior.

DETAILED DESCRIPTION:
Teenage mothers are asked to participate in the study and then randomized into an intervention or control group. Both groups take a multiple choice survey and then are randomized to either watch a video about FAS or not. After the video (or not for the controls) they then take a post video short answer survey. The survey results are then scored and statistical analysis performed to determine whether the video intervention increased their knowledge about FAS and their likelihood to drink alcohol during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant teens aged 12 to 16 years

Exclusion Criteria:

Ages: 12 Years to 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2006-05; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To determine whether an educational video on FAS increases maternal knowledge on the subject and affects their likelihood to drink alcohol. | Immediate

CONTACTS AND LOCATIONS:
Overall Officials: Tammy Camp, MD, Principal Investigator — Texas Tech Department of Pediatrics
Locations (1):
- Grand Expectations, Lubbock, Texas, United States